CLINICAL TRIAL: NCT06266351
Title: EVALUATION of CATS TONOMETER PRISM in LASIK SUBJECTS
Status: Completed | Type: Observational
Sponsor: Intuor Technologies, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: LASIKIOP
Record Dates: First submitted 2024-02-11; First posted 2024-02-20 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-02

CONDITIONS: Glaucoma; Ocular Hypertension; Normal Tension Glaucoma
MeSH Terms: conditions — Glaucoma; Ocular Hypertension; Low Tension Glaucoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- IOP measurement with CATS
  Interventions: Device: This is observational IOP measurement
- IOP measurement with GAT
  Interventions: Device: This is observational IOP measurement

INTERVENTIONS:
Device: This is observational IOP measurement — IOP measurement of patients having LASIK with both CATS and GAT

SUMMARY:
The CATS Tonometer prism clinical study is intended to determine repeatability of intraocular pressure measurement in human corneas which have undergone a LASIK procedure when compared to a standard Goldmann prism, validating the human LASIK eye findings comparing CATS Tonometer and Goldmann prisms to intracameral pressure in cadaver eyes.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet the following inclusion criteria to be eligible to participate in this clinical trial:

* At least 22 years of age and undergone LASIK treatment
* Subject has a clear understanding, English speakingand agrees to all the conditions of the informed consent form

Exclusion Criteria:

* Subjects will be excluded from participation if they meet the following criteria:

  * Subject has undergone ocular surgery within the last 3 months or LASIK within 6 months
  * Pregnant or nursing women
  * Those who have had previous corneal surgery excluding LASIK
  * Keratoconus
  * Corneal scarring
  * Microphthalmos
  * Buphthalmos
  * Dry eyes with clinical epithelial breakdown upon exam
  * Lid squeezers - blepharospasm
  * Nystagmus
  * Corneal or conjunctival infection.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects must meet the following inclusion criteria to be eligible to participate in this clinical trial:
  * At least 22 years of age and undergone LASIK treatment
  * Subject has a clear understanding, English speakingand agrees to all the conditions of the informed consent form
Sampling Method: Non-Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2024-02-12 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
IOP measurement difference between CATS and GAT in LASIK patients | single measurement 1 day
  IOP measurement

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Arizona Eye Consultants, Tucson, Arizona
  - Eye Specialty Group, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided
likely will provide deindentified data